CLINICAL TRIAL: NCT05705193
Title: Computerized Cognitive Remediation of Long COVID Symptoms in Older Adults
Brief Title: Brain-Training Treatment for Long COVID in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Cutter Lindbergh, Assistant Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-089-2; Departmental Funds (Other: UConn Health); P30AG067988 (NIH)
Record Dates: First submitted 2023-01-26; First posted 2023-01-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19 Syndrome
Keywords: Post-Acute COVID-19 Syndrome; Computerized Cognitive Remediation; Older Adults
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computerized Cognitive Remediation (Experimental)
  Interventions: Other: NeuroFlex (computerized gamified tasks)

INTERVENTIONS:
Other: NeuroFlex (computerized gamified tasks) — The computerized cognitive remediation intervention ("NeuroFlex") consists of a series of gamified tasks (e.g., BrainHQ, Neurogrow, Ultimate Word Master) administered via computer tablet. The intervention provides both "bottom up" training to improve basic processing of sensory stimuli and "top down" training to improve executive functions. Participants will be asked to complete approximately 7.5 hours a week of computer treatment over an approximately 6-week period, for a total of approximately 45 hours of treatment. The treatment will be completed remotely by the participant within their own home or other private location that is most convenient for the participant.

SUMMARY:
This research is being done to collect preliminary data on the potential of computerized "brain-training" exercises for treating Long COVID symptoms in older adults. The investigators hypothesize that computerized brain-training will be an acceptable and feasible intervention for treating Long COVID symptoms in older adults. The investigators also expect to provide initial evidence that computerized brain-training has potential for improving thinking, mood, and other aspects of everyday functioning in older adults with Long COVID.

DETAILED DESCRIPTION:
Some patients who contract coronavirus disease 2019 (COVID-19), especially older adults, show lingering neuropsychiatric symptoms such as cognitive impairment, brain fog, and depression. These neuropsychiatric symptoms-commonly referred to under the umbrella term "Long COVID"-are debilitating and may last for months or even years after viral infection. The purpose of the present study is to help address this public health crisis by determining whether computerized "brain-training" treatment has potential for improving thinking, mood, and other aspects of functioning in older adults with Long COVID. More specifically, the first aim is to determine the acceptability and feasibility of using brain-training treatment in individuals with Long COVID. The second aim is to evaluate for potential efficacy by determining whether brain-training treatment appears to improve cognitive function, mood, and other aspects of daily functioning in Long COVID.

ELIGIBILITY:
Inclusion Criteria:

* prior history of COVID-19 based on Centers for Disease Control and Prevention (CDC) guidelines including a positive laboratory test (e.g., nucleic acid amplification test) or a positive rapid test
* age ≥ 60 years old
* current self-reported cognitive symptoms persisting after the acute phase of the illness (i.e., >4 weeks after COVID-19 symptom onset) that cannot be explained by alternative diagnoses
* evidence of subjective cognitive impairment with a Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) Perceived Cognitive Impairment (PCI) Subscale Score of ≤ 40 and/or endorsing any item on the FACT-Cog PCI Subscale as occurring nearly every day or several times a day
* Telephone Interview for Cognitive Status (TICS) ≥ 27
* fluent in English
* off psychiatric medications or on a stable dose for at least 1 month prior to commencing the study with no intention to change dose prior to completion of the study.

Exclusion Criteria:

* history of neurological disorder or other medical condition with potential to impair cognitive functioning or interfere with study participation (e.g., epilepsy, stroke, dementia, head trauma followed by persistent neurological deficits or known structural brain abnormalities)
* prior diagnosis of Mild Cognitive Impairment (MCI) or Mild Neurocognitive Disorder unrelated to the participant's history of COVID-19
* history of significant psychiatric illness per Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), criteria that may interfere with study participation or confound results (e.g., schizophrenia or other psychotic disorder, bipolar and related disorders, major depressive disorder with psychotic features, personality disorder)
* history of significant neurodevelopmental condition that may interfere with study participation or confound results (e.g., intellectual disability, autism spectrum disorder)
* alcohol or other substance use disorder within the past 2 years
* significant sensory or motor impairments (e.g., blindness) that may interfere with the ability to complete neuropsychological measures or engage in the intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Treatment Acceptability/Adherence Scale (TAAS) | The investigators will evaluate TAAS Total Score at the outset of treatment (expected/anticipated acceptability and adherence) and at post-treatment (6 weeks)
  Treatment acceptability and adherence as measured by the TAAS Total Score; higher scores on this self-report measure indicate greater treatment acceptability and adherence
Credibility/Expectancy Questionnaire (CEQ) | The investigators will evaluate CEQ Total Score at the outset of treatment (to assess initial perceptions of treatment credibility) and at post-treatment (6 weeks)
  Treatment credibility and expectancy as measured by the CEQ Total Score; higher scores on this self-report measure indicate greater treatment credibility and expectancy
System Usability Scale (SUS) | The investigators will evaluate SUS Total Score at the outset of treatment (to assess initial perceptions of treatment usability) and at post-treatment (6 weeks)
  Usability of the intervention as measured by the SUS Total Score; higher scores on this self-report measure indicate greater perceived usability
Feasibility (proportion of subjects who agree to participate in the offered treatment, complete assigned exercises, and complete the entire treatment regimen) | Our feasibility criteria will be assessed by calculating percentages at the conclusion of the study
  Feasibility will be assessed according to the following criteria: 1) at least 80% of eligible subjects offered the treatment agree to participate; 2) subjects will complete at least 80% of assigned treatment exercises; 3) at least 80% of participants who start the treatment will finish it.

SECONDARY OUTCOMES:
Trail Making Test Part B | The investigators will evaluate change in time (seconds) to complete the Trail Making Test Part B at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Set-shifting abilities as measured by time to complete the Trail Making Test Part B in seconds; lower scores indicate better set-shifting performance
Montgomery-Asberg Depression Scale (MADRS) | The investigators will evaluate change in Total MADRS Score at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Depressive symptoms as measured by the Total MADRS Score; lower scores indicate less depressive symptoms
World Health Organization Disability Assessment Schedule (WHODAS) | The investigators will evaluate change in Total WHODAS Score at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Functional disability as measured by the Total WHODAS Score; lower scores indicate less functional disability
Everyday Cognition (ECog) | The investigators will evaluate change in Total ECog Score at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Subjective cognitive concerns as measured by the Total ECog Score; lower scores indicate less subjective cognitive concern
Verbal Fluency | The investigators will evaluate change in total number of words produced at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Verbal generativity as measured by the total number of words produced according to pre-specified rules; higher scores indicate better verbal generativity performance
Stroop Color and Word Test | The investigators will evaluate change in total correct responses at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Inhibitory control as measured by total correct responses on the inhibition condition of the Stroop Test; higher scores indicate better inhibitory control performance
Fatigue Assessment Scale (FAS) | The investigators will evaluate change in total FAS Score at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Fatigue as measured by the Total FAS Score; lower scores indicate less fatigue
California Verbal Learning Test (CVLT) | The investigators will evaluate change in long delayed free recall at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Verbal memory as measured by the total number of words correctly recalled on the long delayed free recall trial; higher scores indicate better episodic memory performance
Short Physical Performance Battery (SPPB) | The investigators will evaluate change in physical performance at post-treatment (6 weeks) relative to pre-treatment (baseline)
  Physical performance as measured by the Total SPPB Score; higher scores indicate better physical performance.

CONTACTS AND LOCATIONS:
Overall Officials: Cutter Lindbergh, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No